CLINICAL TRIAL: NCT04873167
Title: Effects of Adherence to a Mediterranean Diet Style on Cardiovascular Risk by Means Its Influence on Serum Levels of Ceramides and on Some Atherothrombotic Candidate Gene Expression
Brief Title: Effects of Adherence to a Mediterranean Diet Style on Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Antonino Tuttolomondo, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U Palermo
Record Dates: First submitted 2021-04-17; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Diet, Fat-Restricted; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Fat Diet (Experimental): subjects subjected to a low-fat dietary regime
  Interventions: Behavioral: low fat
- Mediterranean Diet (Experimental): subjects subjected to a mediterranean dietary regime
  Interventions: Behavioral: mediterranean diet

INTERVENTIONS:
Behavioral: low fat — subjects subjected to a low-fat dietary regime
  Arms: Low Fat Diet
Behavioral: mediterranean diet — subjects subjected to a mediterranean dietary regime
  Arms: Mediterranean Diet

SUMMARY:
Evaluation of the effect of adherence to Mediterranean Diet on some surrogate vascular markers and on gene expression of some cardiometabolic genes

DETAILED DESCRIPTION:
The investigators have designed a study project to evaluate in a sample of patients with high cardiovascular risk:

1. The effects of adherence to Mediterranean Diet on serum levels of some metabolic variables (glucose blood levels, serum LDL cholesterol, serum total cholesterol, serum triglycerides)
2. The effects of adherence to Mediterranean Diet on serum levels of some ceramides and of adiponectin and resistin at 6 and 12-month follow-up
3. The effects of adherence to a Mediterranean Diet style on some surrogate markers of vascular damage such ad endothelial function measured by means of the evaluation of reactive hyperemia index (RHI) and arterial stiffness markers (PWV, AIX) at 6 and 12-month follow-ups
4. The effects of adherence to Mediterranean Diet on the genetic expression of some cardiometabolic and atherothrombotic candidate genes at 12-month follow-up
5. The effects of the Mediterranean diet adherence on the incidence of cardio and cerebrovascular events at 12 and 18 month follow-ups considering respectively:

   1. composite endpoint: myocardial infarction, ischemic stroke and death from cardiovascular causes
   2. secondary endpoint: myocardial infarction, stroke, death from cardiovascular causes

ELIGIBILITY:
Inclusion Criteria:

* at least two of the following eligibility criteria:

  1. Type 2 diabetes mellitus
  2. Arterial hypertension
  3. BMI ≥ 25
  4. Active smoking
  5. Family history of early cardiovascular disease
  6. Previous cardiovascular or cerebrovascular events (> 6 months)

Exclusion Criteria:

* All patients with recent (<6 months) cardiovascular or cerebrovascular events were excluded.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Effects on metabolic variables | Baseline to 12 months
  Effects of adherence to Mediterranean Diet in determining a change in serum levels of some metabolic variables (glucose blood levels in mg/dl, serum LDL cholesterol in mg/dl, serum Total cholesterol in mg/dl, serum triglycerides in mg/dl) from baseline to 12 months.

SECONDARY OUTCOMES:
effects on serum resistin serum levels | Baseline to 12 months
  Effects of adherence to Mediterranean Diet in determining a change from baseline serum levels of resistin in ng/ml to 6 and 12 month follow-ups.
effects on serum ceramides. | Baseline to 12 months
  Effects of adherence to Mediterranean Diet in determining a change from baseline serum levels of some ceramides in ug/ml to 6 and 12 month follow-ups.
effects on adiponectin serum levels | Baseline to 12 months
  Effects of adherence to Mediterranean Diet in determining a change from baseline serum levels of adiponectin in mcg/ml to 6 and 12 month follow-ups.
Effects on surrogate cardiovascular marker (endothelial dysfunction) | Baseline to 12 months
  Effects of adherence to a Mediterranean Diet style in determining a change from baseline values of some surrogate markers of vascular damage such as endothelial function measured by means the evaluation of RHI (reactive hyperemia index) to 6 and 12 month follow-ups
Effects on arterial stiffness indexes | Baseline to 12 months
  Effects of adherence to a Mediterranean Diet style in determining a change from baseline values of some surrogate markers of vascular damage such as arterial stiffness markers (PWV in m/s, AIX in 100 × ((P2-P1)/(Pulse Pressure) to 6 and 12 month follow-ups
effects on gene expression | Baseline and12 months
  Effects of adherence to Mediterranean Diet in determining a change in the genetic expression of some cardiometabolic and atherothrombotic candidate genes (- C_29347861_10, rs7903146, SNP (single nucleotide polymorphism) of TCF7L2 (Transcription Factor 7 Like 2)
  * C_32667060_10, rs17782313, by MC4R ( melanocortin receptor 4)
  * C_30090620_10, rs9939609, SNP of FTO (Fat mass and obesity-associated protein)
  * C_29347861_10, rs7903146, SNP of TCF7L2
  * C_9639448_10, rs13702, SNP of LPL (lipoprotein lipase) ) at 12 month follow-up with Real-Time PCR (polymerase chain reaction assay)
Effects on cardiovascular events | Baseline to 24 months
  Effects of the Mediterranean diet adherence on the incidence of new cardio and cerebrovascular events at 12 and 24 months follow ups considering a composite endpoint: myocardial infarction, ischemic stroke and death from cardiovascular causes.

CONTACTS AND LOCATIONS:
Overall Officials: Antonino tuttolomondo, Principal Investigator — University of Palermo
Locations (1):
- University of Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daidone M, Casuccio A, Puleo MG, Del Cuore A, Pacinella G, Di Chiara T, Di Raimondo D, Immordino P, Tuttolomondo A. Mediterranean diet effects on vascular health and serum levels of adipokines and ceramides. PLoS One. 2024 May 29;19(5):e0300844. doi: 10.1371/journal.pone.0300844. eCollection 2024. PMID 38809909